CLINICAL TRIAL: NCT03770754
Title: Instrumentation Time Efficiency and Histologically the Debriding Efficacy of Rotary and Hand Instrumentation Performed on Human Primary Teeth.
Brief Title: Instrumentation Time Efficiency and Histologically the Debriding Efficacy.
Acronym: ITE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Principal Investigator, Jorge Paredes Vieyra, Chairman of Post graduate Programs in Dentistry, Universidad Autonoma de Baja California
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Intrumentation time efficiency
Record Dates: First submitted 2018-11-20; First posted 2018-12-10 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Necrosis
Keywords: clean; Primary Root canal; rotary instrumentation
MeSH Terms: conditions — Necrosis

STUDY DESIGN:
Intervention Model Description: All clinical procedures and measurements were conducted by the author. A #0 periapical radiograph was taken for each tooth in buccolingual projection to allow proper selection. The selected teeth included 7 second maxillary molars (three canals each), 9 first maxillary molars (2 canals each), 3 central incisors (one canal each), 18 first mandibular molars (2 canals each), 8 second mandibular molars (three canals each) for a total of 45 teeth with 102 canals (Table 1).
  A standard session time recommended by the pedodontists was approximately 20-35 minutes in length to allow for acceptable time for completion of treatment. All treatment was performed by the author. As a novel treatment in Pedodontics, were included electronic apex locator (EAL), EndoVac system and two rotary systems: LightSpeed LSX instruments and ProTaper Next.
Who Masked: Participant, Investigator
Masking Description: Certified endodontists trained in the procedures, devices, and systems investigated took part in the research. All experts tracked a pre-established procedure for Rotary instrument systems and Endo vac system.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Experimental): Control Group (n= 15): the root canals were prepared manually with K-files (Dentsply-Maillefer, Ballaigues, Switzerland) and "step back technique" up to size #35.
  Interventions: Procedure: Clean and shape Control group; Procedure: Cleand and shape Group 1; Procedure: Clean and shape Group 2
- Group 1 (Experimental): Group 1 (n= 15): the root canals were instrumented with rotary LightSpeed LSX instruments (Discus Dental, Culver City, CA, USA). They were used to complete the canal preparation to a size #50 for the anteriors and molar teeth to size #40.
  Interventions: Procedure: Clean and shape Control group; Procedure: Cleand and shape Group 1; Procedure: Clean and shape Group 2
- Group 2 (Experimental): Group 2 (n= 15): root canals were instrumented with ProTaper Next (Dentsply Maillefer, Ballaigues, Switzerland) using X1, X2 to X3. 0.5% NaOCl was used for irrigation.
  Interventions: Procedure: Clean and shape Control group; Procedure: Cleand and shape Group 1; Procedure: Clean and shape Group 2

INTERVENTIONS:
Procedure: Clean and shape Control group — For the control group the root canals were prepared manually with K-files and "step back technique" up to size #35. For this group were administered Tylenol
Procedure: Cleand and shape Group 1 — For the Group 1, LightSpeed LSX rotary instruments (Discus Dental, Culver City, CA, USA) were used to complete the canal preparation to a size #50 for the anteriors and molars to size #40. After procedures were administered Tylenol
Procedure: Clean and shape Group 2 — For the group 2 the root canals were instrumented with ProTaper ﬁles using X1, X2 (21mm) to X3 (21mm). 0.5% NaOCl was used for irrigation, the original protocol suggested by ProTaper for permanent teeth was simplified for this study.
  After clinical procedures Tylenol were administered

SUMMARY:
The goal of pulp therapy in the primary dentition is to retain the primary tooth as a fully functional part of the dentition, allowing at the same time for mastication, phonation, swallowing, and the preservation of the space required for the eruption of the permanent tooth. The premature loss of primary teeth may cause changes in the chronology and sequence of eruption of permanent teeth. Maintenance of primary teeth until physiological exfoliation prevents deleterious habits in children.

The primary objectives of cleaning and shaping the root canal system are removing soft and hard tissue containing bacteria, providing a path for irrigants to the apical third, supplying space for medicaments and subsequent obturation, retaining the integrity of radicular structure. The choice between pulpotomy and pulpectomy is generally based on the severity of the symptoms clinically and/or radiographically. When indicated, the primary tooth pulpotomy is a relatively simple procedure with generally good clinical results.

DETAILED DESCRIPTION:
Patient selection was based on the following criteria:

* the aims and requirements of the study were freely accepted by the parents;
* primary molars with at least 11.0 ± 1.0 mm of working length
* Treatment was limited to patients in good health;
* All teeth had vital and non-vital pulps without a sinus tract;
* Excess of bleeding during a pulpotomy; 6) Presence of enough coronal tooth and root structure;
* No prior pulpectomy treatment on the involved tooth,
* absence of perforation in the internal and/or external furcation area and
* No analgesics or antibiotics were used before the clinical procedures began. Exclusion criteria were patients without inclusion requirements or failure to obtain parent´s authorization, and were excluded if they were older than 7 years old, had a positive history of antibiotic use within the past month, diabetic, hemophilic or if the tooth had root resorption or been previously accessed and initiated a pulpectomy.

Once eligibility was conﬁrmed, the parents were informed of the study design, the clinical procedure involved, and the associated risks. Patients aged 4-7 years of age were enrolled in this study, forty-five teeth (19 maxillaries and 26 mandibular teeth), which had a total of 102 canals and completely formed apices and of minimum 10 mm root length were selected. All selected teeth had mature apexes with no radiographic sign of root resorption.

Of the 45 treated primary molars, 31 teeth were diagnosed as having chronic pulpitis, and 14 as having pulp necrosis that responded negative to hot and cold tests; and, clinically, all pulps were conﬁrmed to be necrotic on entrance into the pulp chamber. Informed consent was obtained and written by the parents from each patient in accordance with the approval of the study by the ethical board of the Universidad Autónoma de Baja California, Facultad de Odontología Tijuana, México. All clinical procedures and measurements were conducted by the author.

A #0 periapical radiograph was taken for each tooth in buccolingual projection to allow proper selection. The selected teeth included 7 second maxillary molars (three canals each), 9 first maxillary molars (2 canals each), 3 central incisors (one canal each), 18 first mandibular molars (2 canals each), 8 second mandibular molars (three canals each) for a total of 45 teeth with 102 canals.

A standard session time recommended by the pedodontists was approximately 20-35 minutes in length to allow for acceptable time for completion of treatment. All treatment was performed by the author. As a novel treatment in Pedodontics, were included electronic apex locator (EAL), EndoVac system and two rotary systems: LightSpeed LSX instruments and ProTaper Next.

The teeth were randomly divided into 3 groups (each tooth was considered as an experimental unit): Control Group (n= 15): the root canals were prepared manually with K-files (Dentsply-Maillefer, Ballaigues, Switzerland) and "step back technique" up to size #35.

Group 1 (n= 15): the root canals were instrumented with rotary LightSpeed LSX instruments (Discus Dental, Culver City, CA, USA). They were used to complete the canal preparation to a size #50 for the anteriors and molar teeth to size #40.

Group 2 (n= 15): root canals were instrumented with ProTaper Next (Dentsply Maillefer, Ballaigues, Switzerland) using X1, X2 to X3. 0.5% NaOCl was used for irrigation. The instrumentation time was measured for all the procedures and the results were analyzed with student's t-test. All statistical procedures were computed with SPSS 21.0 (SPSS Inc., Chicago, IL, USA). The Student t test was used to compare data whether there were statistically signiﬁcant differences between the results obtained clinically. Signiﬁcance was set at p < 0.05.

Pilot study. All the procedures were done in extracted primary teeth, they were prepared and disinfected before using the instgruments. After the debridement of the canals, the teeth were sectioned longitudinally and observed under microscope.

Clinical Protocol. After local anesthesia by 2% lidocaine with 1:100,000 epinephrine (58 Rue du Pont de Creteil, Saint - Maur des Fossés F-94100, France) and rubber dam isolation the tooth was disinfected with 2.5% NaOCl (Ultra bleach, Bentonville, AR, USA).

All caries was removed and endodontic access cavities made with sterile high speed carbide # 331 (SS White. Lakewood, NJ). The cervical third of each canal was ﬂared with a SX ProTaper ﬁle (Maillefer, Ballaigues, Switzerland).

Each canal was irrigated consequently with 2.0 cc 0.5% sodium hypochlorite. The final rinse was aspirated but no attempt was made to dry the canals. Working length was established with the Root ZX Electronic Apex Locator (J Morita, Irvine, CA) and confirmed radiographically. The canals were negotiated and enlarged with K-files hand instruments (Dentsply-Maillefer, Ballaigues, Switzerland) until reaching an ISO #20 at the working length.

The Root ZX was used in accordance with the manufacturer's instructions. The buccal clip was attached to the patient's lip, and the probe was connected to a stainless steel 15 K-ﬁle. The ﬁle was advanced within the root canal to a point just beyond the major foramen, as indicated by the ﬂashing APEX bar on the liquid crystal display of the EAL.

When the file was in position the LCD display showed a ﬂashing bar between APEX and 1. Measurements were considered to be correct if the instrument remained constant for at least 4-5 seconds. A digital photograph was taken and stored in Adobe Photoshop 5.5 (Adobe Systems Inc., San Jose, CA, USA). The position of the file tip for each root canal were evaluated by two examiners, if the two examiners disagreed a third previously calibrated researcher was asked to make the ﬁnal decision. The ﬁnal WL was established to be 1 mm coronal to the major foramen (12).

For the control group the root canals were prepared manually with K-files and "step back technique" up to size #35. For the Group 1, LightSpeed LSX rotary instruments (Discus Dental, Culver City, CA, USA) were used to complete the canal preparation to a size #50 for the anteriors and molars to size #40.

For the group 2 the root canals were instrumented with ProTaper ﬁles using X1, X2 (21mm) to X3 (21mm). 0.5% NaOCl was used for irrigation, the original protocol suggested by ProTaper for permanent teeth was simplified for this study.

After completion of canal instrumentation, all canals were irrigated with distilled water for 30 seconds using the EndoVac irrigation system (Discus Dental, Culver City, CA, USA).

The EndoVac system is able to apply the irrigant to working length and evacuate it using apical negative pressure. The negative pressure avoids forcing the irrigant beyond the apex into the periapical tissues.

The canals were dried with sterile paper points and obturated at the same appointment using calcium hydroxide and iodoform paste (Pearson Dental, Sylmar CA) by using pluggers or syringes (Messing Root Canal Gun, PD, Vevey, Switzerland). Access cavities of anterior teeth were etched and restored with Fuji IX (GC Corp, Tokyo, Japan). For posterior teeth, a buildup restoration was placed by using the same etching technique and Fuji IX or temporary metallic crown.

A stopwatch with alarm (http://stopwatch.onlineclock.net/) was used to record instrumentation time for each group.

Children were recalled for clinical and radiographic examinations were evaluated, based on the criteria of Coll and Sadrian at 6-month intervals for a follow-up period of 2 years. Teeth that exhibited no symptoms of pain, tenderness to percussion, swelling, sinus tract, or pathological mobility were judged clinically successful (42 teeth).

Teeth that showed no evidence of periradicular or interradicular radiolucency, internal or external root resorption, or periodontal ligament space widening were judged raiographically successful. Radiographic evidence of pulp canal obliteration was noted, but it was not regarded as failure.

ELIGIBILITY:
Inclusion Criteria:

* the aims and requirements of the study were freely accepted by the parents
* primary molars with at least 11.0 ± 1.0 mm of working length
* Treatment was limited to patients in good health;
* All teeth had vital and non-vital pulps without a sinus tract;
* Excess of bleeding during a pulpotomy;
* Presence of enough coronal tooth and root structure;
* No prior pulpectomy treatment on the involved tooth,
* absence of perforation in the internal and/or external furcation area and
* No analgesics or antibiotics were used before the clinical procedures began.

Exclusion Criteria:

* patients without inclusion requirements or failure to obtain parent´s authorization, .) patients older than 7 years old,
* had a positive history of antibiotic use within the past month,
* diabetic, hemophilic
* if the tooth had root resorption or been previously accessed and initiated a pulpectomy.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-09-20 (Estimated)

PRIMARY OUTCOMES:
Clinical Success | clean and shape with a scale and an average of 3 weeks
  Defined as teeth that exhibited no symptoms of pain, tenderness to percussion, swelling, sinus tract, or pathological mobility

SECONDARY OUTCOMES:
Radiological success | obtain the evaluation in about 5 days
  Defined as teeth that showed no evidence of periradicular or interradicular radiolucency, internal or external root resorption, or periodontal ligament space widening

CONTACTS AND LOCATIONS:
Locations (4):
- Mexico (4):
  - Jorge Paredes Vieyra, Tijuana, Baja Califronia
  - Jorge Paredes Vieyra, Tijuana, Estado de Baja California
  - Jose Clemente Orozco, Tijuana, Estado de Baja California
  - Jose Clemente, Tijuana, Estado de Baja California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paredes-Vieyra J, Enriquez FJ. Success rate of single- versus two-visit root canal treatment of teeth with apical periodontitis: a randomized controlled trial. J Endod. 2012 Sep;38(9):1164-9. doi: 10.1016/j.joen.2012.05.021. Epub 2012 Jul 26. PMID 22892729